CLINICAL TRIAL: NCT05287646
Title: Quantifying Bone and Skin Movement in the Residual Limb-Socket Interface of Individuals With Transtibial Amputation Using Dynamic Stereo X-Ray
Brief Title: Quantifying Bone and Skin Movement in the Residual Limb of Individuals With Transtibial Amputation Using Dynamic Stereo X-Ray
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Rutgers University (Other); University of Rhode Island (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A3700-R
Record Dates: First submitted 2022-03-09; First posted 2022-03-18 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Amputation, Lower Limb
Keywords: Prosthesis Fitting; Prosthetic Suspension Systems; Dynamic Stereo X-Ray; Biplanar Fluoroscopy; Transtibial Amputation; Pistoning; Elevated Vacuum Suspension; Suction Suspension; Lower Extremity Amputation

STUDY DESIGN:
Intervention Model Description: A randomized, block, cross-over design will be used to evaluate the residual limb-socket fit. A group of 11 (Group 1) and a group of 10 (Group 2) participants will be formed. Participants in Group 1 will first be tested with the elevated vacuum system active and then repeat all procedures with the elevated vacuum system inactive. Participants in Group 2 will first be tested with the elevated vacuum system inactive and then repeat the tasks with the elevated vacuum system active.
Masking Description: The statistician will be masked to the intervention order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Suction Suspension First (Active Comparator): The residual limb will be imaged during dynamic activities while participants use suction suspension first, then while participants use elevated vacuum suspension. Dynamic stereo x-ray will take place 4-weeks after socket fitting.
  Interventions: Device: Suction Suspension First
- Elevated Vacuum Suspension First (Active Comparator): The residual limb will be imaged during dynamic activities while participants use elevated vacuum suspension first, then while participants use suction suspension. Dynamic stereo x-ray will take place 4-weeks after socket fitting.
  Interventions: Device: Elevated Vacuum Suspension First

INTERVENTIONS:
Device: Suction Suspension First — Participants will be fit with a socket capable of being suspended by both traditional suction and elevated vacuum. Participants will be assessed first with the elevated vacuum system inactive (traditional suction). Residual limb kinematics and skin deformation during movement tasks will be evaluated utilizing dynamic stereo x-ray. The evaluation will then be repeated with the elevated vacuum system active.
  Arms: Suction Suspension First
Device: Elevated Vacuum Suspension First — Participants will be fit with a socket capable of being suspended by both traditional suction and elevated vacuum. Participants will be assessed first with the elevated vacuum system active. Residual limb kinematics and skin deformation during movement tasks will be evaluated utilizing dynamic stereo x-ray. The evaluation will then be repeated with the elevated vacuum system inactive.
  Arms: Elevated Vacuum Suspension First

SUMMARY:
Individuals with lower extremity amputation are often challenged by complications that arise from poor prosthetic fit, including movement of the residual limb in the socket, known as pistoning. Pistoning can lead to gait instability, skin problems, and pain. Different prosthetic suspension systems have been developed to decrease this motion, including elevated vacuum suspension, which utilizes a pump to draw air from the socket. However, scientific analyses to understand the movement between the limb and socket have yet to be performed with a high level of accuracy. This study will use a state-of-the art imaging technique, known as dynamic stereo x-ray, to quantify the 3D movement of the residual limb in the socket. It is hypothesized that dynamic stereo x-ray will be a sensitive method to measure differences in residual limb movement between 2 different socket suspension techniques: suction and elevated vacuum suspension. This information is critical for advancing prosthetic treatments to reduce secondary conditions and degenerative changes that result from poor prosthetic fit.

DETAILED DESCRIPTION:
Individuals with lower extremity amputation (LEA) often experience relative motion between their residual limb and the prosthetic socket, such as vertical translation and axial rotation, which can cause inefficient dynamic load transmission from the distal prosthetic components to the residual limb. This can lead to significant secondary consequences, such as pain, gait deviations, and discomfort that limit mobility and autonomy. Assessments of the relative motion between the bone and the prosthetic socket have been performed, but there is little existing data on dynamic, in vivo residual limb-socket kinematics since most investigations have been performed using non-dynamic testing protocols, static measurements, or with unvalidated surface marker-based motion capture systems. Dynamic Stereo X-ray (DSX) is an advanced imaging technology that can quantify 3D bone movement and tissue/liner deformation inside a prosthetic socket during dynamic activities.

There is a substantial gap in our understanding of the complex mechanics of the residual limb-socket interface during dynamic activities that limit the ability to improve prosthetic design. The goals for this project are to develop the analytical tools to quantify both the dynamic, in-vivo kinematics between the residual limb and socket, as well as the mechanism of residual tissue/liner deformation. In order to validate the sensitivity of this methodology to differences in socket suspension, 2 suspension systems will be evaluated: elevated vacuum and traditional suction. It is hypothesized that an efficient and highly accurate method to quantify the dynamic interaction between the residual limb and prosthetic socket will be sensitive enough to distinguish between different types of prosthetic socket suspension, which will further the biomechanical understanding of socket design. To do so, the investigators will address the following aims: (1) To optimize the DSX procedural setup for the accurate tracking of the prosthetic socket, skeletal kinematics, and tissue/liner deformation; (2) To quantify the relative motion between the residual tibia and the prosthetic socket during dynamic activities; and (3) To measure the deformation of the skin and liner in the prosthetic socket during dynamic activities.

Twenty-one participants with transtibial amputation will be fit with a socket capable of being suspended via both elevated vacuum and traditional suction. Participants will undergo a 4-week acclimation period and then be tested at the DSX facility. DSX will be utilized to track skeletal and skin/liner motion under both suspension techniques during 3 dynamic activities: treadmill walking at self-selected speed, fast walking (10% faster), and a step-down movement. The performance of the two suspension techniques (active EV and traditional suction) will be tested by quantifying the 3D bone movement of the residual tibia with respect to the prosthetic socket and quantifying liner and soft tissue deformation at the socket-residuum interface.

By using the analytical tools for a highly accurate, in-vivo assessment of residual limb-socket motion, vital foundational information can be provided to aid in the development of new methods and techniques to enhance prosthetic fit that have the potential to reduce secondary physical comorbidities and degenerative changes that result from complications of poor prosthetic load transmission.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral transtibial amputation (any etiology)
* At least 18 years old
* At least 6-months post-amputation
* Current prosthetic users (at least 6 hours/day)

Exclusion Criteria:

* Unable to ambulate on a treadmill at low to moderate speed
* Inability to tolerate the socket suspensions
* Length of the residual limb prohibits socket fitting, dynamic stereo x-ray data capture, or marker placement
* Mental impairment that impedes study compliance
* Skin conditions (i.e. burns or poor skin coverage) as well as those with severe contractures that prevent prior prosthetic wear
* Severe neuropathy, uncontrolled diabetes, have insensate foot, severe phantom pain, or a significant history of skin ulcers
* Any other significant comorbidity that would interfere with the study
* Severe circulatory problems including peripheral vascular disease and pitting edema
* Cognitive deficits or mental health problems that would limit ability to participate fully in the study protocol
* Women who are pregnant or who plan to become pregnant during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2024-01-05 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Changes in dynamic residual tibia kinematics between suspension techniques | 4 weeks post socket fit
  To evaluate the 6 degree of freedom kinematics of the residual limb within the socket, participants with transtibial amputation will walk on a treadmill at a self-selected speed, at a speed 10% faster than their self-selected speed, and also perform a step-down task from an 18 cm high platform. These movement tasks will be completed under 2 conditions: with the elevated suspension active and with the elevated system inactive (traditional suction). Up to 4 trials of dynamic stereo x-ray will be conducted for each task for each socket condition. For each task, dynamic stereo x-ray data will be collected and analyzed to determine underlying bone movement with respect to the socket. Six degree of freedom residual tibia rotations and translations relative to the prosthetic socket will be measured.
Changes in dynamic skin deformation of the residual limb between suspension techniques | 4 weeks post socket fit
  Radio-opaque markers will be placed on the residual limb in specific patterns. Participants will walk on a treadmill at a self-selected speed, at a speed 10% faster than their self-selected speed, and also perform a step-down task from an 18 cm high platform. These movement tasks will be completed under 2 conditions: with the elevated suspension active and with the elevated system inactive (traditional suction). Up to 4 trials of dynamic stereo x-ray will be conducted for each task for each socket condition. For each task, dynamic stereo x-ray data will be collected and analyzed to determine underlying skin deformation. The radio-opaque markers on the skin will be tracked during the dynamic trials, and their trajectories in the socket coordinate system will define the motion of the skin relative to the socket. Shear, defined as the change in angle between the markers, and compression, defined as the change in distance between markers and a neutral position, will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Maikos, PhD, Principal Investigator — VA NY Harbor Healthcare System, New York, NY
Locations (1):
- VA NY Harbor Healthcare System, New York, NY, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be stored in a curated data repository that makes the data underlying scientific publications discoverable, freely usable, and citable, while promoting openly available research integrated with scholarly literature.
Time Frame: After study completion

REFERENCES:
- [Derived] Paglia DN, Chomack JM, Herlihy DV, Wetterstrand C, Kadkoy Y, Duchnycz R, Kelly P, O'Connor JP, D'Andrea SE, Maikos JT. Mitigation of image distortion during mechanical testing within a dynamic stereo x-ray system. Front Bioeng Biotechnol. 2025 May 19;13:1571639. doi: 10.3389/fbioe.2025.1571639. eCollection 2025. PMID 40458257